CLINICAL TRIAL: NCT03043898
Title: Mapping Sound Propagation Through the Human Lung for Better Diagnosis
Status: Terminated | Type: Observational
Why Stopped: COVID-19
Sponsor: Maximilian Nussbaumer (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Maximilian Nussbaumer, Principal Researcher, University of Cambridge
Organization: University of Cambridge (Other)
Other Study IDs: A093684
Record Dates: First submitted 2017-01-30; First posted 2017-02-06 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Bronchomalacia; Asthma; Lung Neoplasms; Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Bronchomalacia; Asthma; Lung Neoplasms; Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Part A(i) Healthy Volunteers: 50 healthy volunteers. Intervention: Lung sound recording for part A(i) of the study.
  Interventions: Other: Lung sound recording
- Part A(ii) Patients: 100 patients with wheezing and/or crackles due to respiratory disease. Intervention: Lung sound recording for part A(ii) of the study.
  Interventions: Other: Lung sound recording
- Part B(i) 'normal' lung structure: 25 patients who are scheduled to have a Bronchoscopy as part of their standard care and are identified by a medical professional as having a 'normal' lung structure.
  Intervention: Lung sound transmission measurement for part B(i) of the study.
  Interventions: Other: Lung sound transmission measurement
- Part B(ii) 'abnormal' lung structure: 25 patients who are scheduled to have a Bronchoscopy as part of their standard care and are identified by a medical professional as having an 'abnormal' lung structure.
  Intervention: Lung sound transmission measurement for part B(ii) of the study.
  Interventions: Other: Lung sound transmission measurement

INTERVENTIONS:
Other: Lung sound transmission measurement — Sound at chest wall is recorded using a sensor array during the bronchoscopy procedure, while a sound is played down the working channel of the bronchoscope.
  Groups: Part B(i) 'normal' lung structure; Part B(ii) 'abnormal' lung structure
Other: Lung sound recording — Lung sounds are recorded using a sensor array.
  Groups: Part A(i) Healthy Volunteers; Part A(ii) Patients

SUMMARY:
This study investigates the propagation of sound from a source in the chest to the chest wall.

The methodology of the study will be to place a sound source at a known location in the chest and measure the acoustic response on the posterior chest wall with an acoustic sensor array.

The sound source will be created by playing sound down the working channel of a bronchoscope and located anatomically using direct imaging.

Subjects will be selected for the study by asking patients undergoing a bronchoscopy procedure whether they would be willing to take part in the experiment in addition to their standard procedure.

Procedures will take place in the Bronchoscopy Unit at Addenbrooke's hospital in Cambridge. The Unit runs regional speciality clinics in severe chronic obstructive pulmonary disease, asthma, lung cancer, bronchomalacia and interstitial lung disease and has a nationally significant interventional bronchoscopy service.

A subsidiary part of the study (Part A) will collect sound recordings from healthy volunteers and patients with common respiratory diseases using the same acoustic sensor array. This is to create a database of lung sounds and quantify inter-subject variability.

The study will last approximately 30 months.

DETAILED DESCRIPTION:
The study has two parts, A and B. Both parts are observational studies of the sounds heard at the chest as recorded by an acoustic array.

In Part A, healthy volunteers and patients at Addenbrooke's hospital will have the chest sounds at their back recorded using an electronic-stethoscope array. This will be done in a single session lasting approximately 30 minutes. 50 healthy volunteers and 100 patients will be included.

In Part B, 50 patients undergoing a bronchoscopy at Addenbrooke's hospital will have their bronchoscopy extended by 5-10 minutes so that sounds can be played through the working channel of the bronchoscope and recorded by a microphone array at the posterior chest. Part B will investigate 25 patients with structurally 'normal' lungs (for example patients with Chronic Cough) (Part B(i)), and 25 patients with lung disease that has resulted in an 'abnormal' lung structure (Part B(ii)).

The consultant bronchoscopist will assign the patient to the relevant group based on information from their medical history and their CT scan. For Part B of the study an existing CT scan is an inclusion criterion. CT scans will not be carried out specifically for this study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male of Female, aged 18 years or above.
* Part A(i) Healthy volunteer with no history of smoking, recreational drug use or respiratory disease.
* Part A(ii) Patient admitted to Addenbrooke's with a pulmonary disease resulting in crackles and/or wheezes (as diagnosed by a qualified medical practitioner).
* Part B Patient admitted to Addenbrooke's hospital for a bronchoscopy procedure.
* Part B Appropriate recent imaging available: chest CT within 3 months.
* Part B(i) Lung structure deemed 'normal' by pulmonary physician based on CT scan and medical history.
* Part B(i) Lung structure deemed 'abnormal' by pulmonary physician based on CT scan and medical history.

Exclusion Criteria:

* Informed consent is not given.
* Subject is under 18 years old.
* WHO performance status >2.
* Subject is pregnant.
* Subject is unable to understand English.
* Part A(i) History of smoking, recreational drug use or respiratory disease.
* Part A(ii) Condition judged to have no effect on breathing sounds. Patient with crackle or wheeze when quota for crackle or wheeze patients respectively is fulfilled.
* Part B Risk associated with prolonging bronchoscopy procedure judged to be too high by medical professional.
* Part B Appropriate recent imaging (chest CT within 3 months) not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Part A(i) 50 healthy volunteers, taken from the general population.
  Part A(ii) 100 patients, taken from the population of patients at Addenbrooke's Hospital, Cambridge, UK with clear evidence of wheezing and/or crackles due to respiratory disease. We will aim to recruit approximately 50 patients with wheezing and 50 patients with crackles.
  Part B(i) 25 patients, taken from the population of patients on the bronchoscopy list at Addenbrooke's Hospital, Cambridge, UK.
  Part B(ii) 25 patients, taken from the population of patients on the bronchoscopy list at Addenbrooke's Hospital, Cambridge, UK
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Comparison of sound propagation through the human chest in subjects with 'normal' and 'abnormal' lung structure. | Will be assessed when all data for Part B of the study has been collected. Up to 30 months.
  This will use a hypothesis test on features extracted from the time-series array data in Part B of the study.

SECONDARY OUTCOMES:
Database of acoustic response of human chest to a known sound input within the lungs. | Will be assessed when all data for Part B of the study has been collected. Up to 30 months.
  This will consist of acoustic data from an array of acoustic sensors on the posterior back, acoustic data from the sound source, photographs of the back with sensor locations and key anatomical features marked and thorax CT scans. This database will be used to investigate propagation mechanisms and localisation techniques.
Database of lung sound recordings from array on posterior chest. | Will be assessed when all data for Part A of the study has been collected. Up to 30 months.
  This will consist of acoustic data from an array of acoustic sensors at the posterior chest of supine participants taken while these perform a series of breathing exercises. The database will also include basic biometric data.

CONTACTS AND LOCATIONS:
Overall Officials: Pasupathy Sivasothy, PhD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals and the University of Cambridge, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable patient data will be used in publications and made available on the University of Cambridge's data repository DSpace when the results of the study are published.